CLINICAL TRIAL: NCT03713957
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Tolerability of GRF6021 Infusions in Subjects With Parkinson's Disease and Cognitive Impairment
Brief Title: A Study to Assess the Safety of GRF6021 Infusions in Subjects With Parkinson's Disease and Cognitive Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkahest, Inc. (Industry)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Alkahest study 6021-201
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Parkinson Disease
Keywords: Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders; Parkinson's Disease; Dementia
MeSH Terms: conditions — Parkinson Disease; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders; Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GRF6021 (Experimental): Subjects will receive GRF6021 for 5 consecutive days at Week 1 and Week 13.
  Interventions: Drug: GRF6021
- Placebo (Placebo Comparator): Subjects will receive Placebo for 5 consecutive days at Week 1 and Week 13.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GRF6021 — GRF6021 for IV infusion
  Arms: GRF6021
Other: Placebo — Placebo for IV infusion
  Arms: Placebo

SUMMARY:
This study will evaluate the safety, tolerability, and potential effects on cognition of GRF6021, a plasma-derived product, administered as an intravenous (IV) infusion, to subjects with Parkinson's disease and cognitive impairment.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to assess the safety and tolerability of GRF6021, a plasma derived product, administered by intravenous (IV) infusion to subjects with Parkinson's disease (PD) and cognitive impairment. The study duration for the subjects will be approximately 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease (PD), with at least 1 year of PD symptoms.
* Diagnosis of PD with mild cognitive impairment (PD-MCI) or probable or possible Parkinson's disease dementia according to Movement Disorder Society's Clinical Diagnostic criteria.
* Score on the Montreal Cognitive Assessment (MoCA) of 13-25.
* Modified Hoehn and Yahr Stages 1-4.
* Modified Hachinski Ischemic Scale (MHIS) score of 4 or less.

Exclusion Criteria:

* History of blood coagulation disorders or hypercoagulability.
* Current use of anticoagulant therapy. Use of antiplatelet drugs (e.g., aspirin or clopidogrel) is acceptable.
* Prior hypersensitivity reaction to any human blood product or any IV infusion.
* Treatment with any human blood product, including transfusions and IV immunoglobulin, during the 6 months prior to screening.
* History of immunoglobulin A or haptoglobin deficiency; stroke, anaphylaxis, or thromboembolic complications of IV immunoglobulins.
* Heart disease, as evidenced by myocardial infarction, unstable, new onset or severe angina, or congestive heart failure in the 6 months prior to dosing
* Hemoglobin < 10 g/dL in women and < 11 g/dL in men.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkahest Medical Monitor, Study Director — Alkahest, Inc.
Locations (29):
- United States (19):
  - Clinical Trials, Inc., Little Rock, Arkansas
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - Moonshine Research Center, Doral, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - MD Clinical, Hallandale, Florida
  - Research Centers of America, LLC, Hollywood, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Qps_Mra, Llc, South Miami, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - NeuroTrials Research Inc., Atlanta, Georgia
  - Quest Research Institute, Farmington Hills, Michigan
  - SRI Biosciences, Plymouth, Michigan
  - PsychCare Consultants Research, St Louis, Missouri
  - Wake Research, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - UT Southwestern Medical Center, Dallas, Texas
  - Centex Studies, INC., Houston, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
- Alfred Hospital, Melbourne, Victoria, Australia
- France (9):
  - Hopital Neurologique, Bron
  - Hopital Henri Mondor, Créteil
  - CHU Grenoble Alpes, Grenoble
  - Hopital Roger Salengro, Lille
  - Hopital de la Timone, Marseille
  - CHU Caremeau, Nîmes
  - CHU de Poitiers, Poitiers
  - CHU Charles Nicolle, Rouen
  - CHU Purpan - Hopital Pierre Paul Riquet, Toulouse

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GRF6021 | Placebo
Started | 53 | 26
Completed | 35 | 16
Not Completed | 18 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GRF6021 | Placebo | Total
Number analyzed (Participants) | 53 | 26 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (7.63) | 68.4 (8.88) | 67.5 (8.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 26
  Male | 37 | 16 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 13 | 38
  Not Hispanic or Latino | 28 | 13 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 2 | 11
  White | 44 | 24 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47 | 23 | 70
  Australia | 1 | 0 | 1
  France | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Treatment-emergent adverse events identified by MedDRA preferred term and grouped by MedDRA System Organ Class
Time Frame: Approximately 24 Months
Population: The Safety Set includes all subjects at least one dose of the study agent. All safety analyses were performed using the Safety Set, based on treatment received.
Measure: Number; unit: participants
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 51 | 25
participants
  Participants with at least one TEAE | 45 | 20
  Participants with at least one SAE | 5 | 0

2. Secondary Outcome: The Montreal Cognitive Assessment (MoCA) Score.
Description: Change from baseline in the The Montreal Cognitive Assessment (MoCA). The MoCA is a 30-point test, which assess the attention and concentration, executive functions, memory, visuospatial abilities, language abilities, conceptual thinking, calculations, and orientation. Higher scores indicate better cognitive function; the total possible score is 30 and a score of 26 or more is considered normal. A positive value of change means an improvement, and a negative value of change means deterioration. Score range [0 (min) - 30 (Max)].
Time Frame: Change from Baseline to Week 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 44 | 22
score on a scale | 1.30 (3.62) | 0.80 (3.13)

3. Secondary Outcome: Continuity of Attention, Reaction Time Variability, Working Memory, and Episodic Memory on the Cognitive Drug Research Computerized Cognition Battery (CDR-CCB) as Assessed by Change From Baseline in CDR-CCB.
Description: The CDR-CCB is an automated cognitive function assessment system. The secondary efficacy outcomes involved the following composite scores:
  * Continuity of Attention: Min: - 20 # ; 35 #
  * Reaction Time Variability: Min: 0 #; Max: 900 #
  * Quality of Working Memory: Min : 0 # ; Max: 2 #
  * Quality of Episodic Memory: Min: -400 #; Max: 400 #
  Note: # denotes "no specific unit"
  Lower scores reflect poorer ability for Continuity of Attention, Quality of Working Memory, and Quality of Episodic Memory; thus, a negative change from baseline reflects impairment compared to baseline. Whereas, for Reaction Time Variability, higher scores reflect poorer ability, and a positive change from baseline reflects impairment compared to baseline.
Time Frame: Change from Baseline to Week 20
Population: A subset of the Evaluable set comprised of subjects who receive all 10 planned doses, who complete Visit 18 and Visit 19 in window, and who do not have any of the deviations listed below or any other deviation that could potentially affect the assessment of efficacy identified prior to database lock.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 35 | 16
score on a scale
  Continuity of Attention | -0.42 (1.12) | -0.28 (1.12)
  Reaction Time Variability | 4.67 (8.40) | 2.87 (8.40)
  Quality of Working Memory: number analyzed (Participants) | 34 | 16
  Quality of Working Memory | 0.09 (0.12) | -0.04 (0.12)
  Quality of Episodic Memory: number analyzed (Participants) | 33 | 16
  Quality of Episodic Memory | -10.02 (15.82) | 8.65 (15.82)

4. Secondary Outcome: The Delis-Kaplan Executive Function System (D-KEFS) Verbal Fluency.
Description: Change from baseline in the Delis-Kaplan Executive Function System (D-KEFS). The D-KEFS Verbal Fluency test is used for assessment of executive function and has three conditions: Letter Fluency, Category Fluency, and Category Switching. Higher scores indicate more correct responses. A positive value of change means an improvement and a negative value of change means deterioration. The minimum score is 0 and there is no concrete maximum score.
Time Frame: Change from Baseline to Week 20
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 40 | 20
score on a scale | 5.00 [-3.12 to 13.13] | -1.59 [-11.77 to 8.58]

5. Secondary Outcome: The Movement Disorder Society's Unified Parkinson's Disease Rating Scale (MDS-UPDRS) 1, 2, 3, and Total Score.
Description: Change from baseline in the Movement Disorder Society's Unified Parkinson's Disease Rating Scale (MDS-UPDRS). The MDS-UPDRS contains 4 subscales: Part 1, Mentation, Behavior, and Mood; Part 2, Activities of Daily Living; Part 3, Motor; Part 4, Complications nonmotor experiences of daily living (13 items), motor experiences of daily living (13 items), motor examination (18 items), and motor complications (six items). The rating for each item is from 0 (normal) to 4 (severe). The total score for each Part is obtained from the sum of the corresponding item scores. For this study, Parts 1-3 will be completed. Part 1 score ranges from 0 to 52. Part 2 score ranges from 0 to 52. Part 3 score ranges from 0 to 132. Total score possible is 0 to 236.
Time Frame: Change from Baseline to Week 16
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 44 | 22
score on a scale | -8.89 [-13.74 to -4.04] | -9.53 [-16.43 to -2.64]

6. Secondary Outcome: The Schwab and England Activities of Daily Living (SE-ADL) Scale.
Description: Change from baseline in the Schwab and England Activities of Daily Living (SE-ADL). The SE-ADL evaluates patients' perceptions of global functional capacity and dependence. Scoring is expressed in terms of percentage, in 10 steps from 100 to 0 (100%, normal status; 0%, bedridden with vegetative dysfunction), so that the lower the score, the worse the functional status. The range is 0% to 100%.
Time Frame: Change from Baseline to Week 24
Population: The difference between the Number Analyzed at Baseline and week 24 timepoint is due the withdrawal of participants or missed assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 50 | 25
Participants
  Baseline: 100% Independency | 2 | 2
  Baseline: 90% Independency | 10 | 2
  Baseline: 80% Independency | 21 | 11
  Baseline: 70% Independency | 9 | 4
  Baseline: 60% Independency | 3 | 4
  Baseline: 50% Independency | 1 | 0
  Baseline: 40% Independency | 1 | 1
  Baseline: 30% Independency | 3 | 0
  Baseline: 20% Independency | 0 | 1
  Baseline: 10% Independency | 0 | 0
  Baseline: 0% Independency | 0 | 0
  Week 24: number analyzed (Participants) | 43 | 21
  Week 24: 100% Independency | 2 | 1
  Week 24: 90% Independency | 10 | 4
  Week 24: 80% Independency | 15 | 7
  Week 24: 70% Independency | 6 | 4
  Week 24: 60% Independency | 4 | 2
  Week 24: 50% Independency | 3 | 1
  Week 24: 40% Independency | 1 | 0
  Week 24: 30% Independency | 1 | 1
  Week 24: 20% Independency | 0 | 1
  Week 24: 10% Independency | 1 | 0
  Week 24: 0% Independency | 0 | 0

7. Secondary Outcome: The Clinical Impression of Severity Index - PD (CISI-PD).
Description: Change from baseline in The Clinical Impression of Severity Index PD (CISI-PD). The CISI-PD is a severity index formed by four items (motor signs, disability, motor complications, and cognitive status), rated 0 (not at all) to 6 (very severe or completely disabled); the possible scores range from 0 to 24. A total score is calculated by summing the item scores. Higher scores indicate worse severity. A negative value of change means an improvement and a positive value of change means deterioration.
Time Frame: Change from Baseline to Week 24
Measure: Least Squares Mean (95% Confidence Interval); unit: change from baseline score
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 43 | 21
change from baseline score | -0.54 [-1.91 to 0.83] | -0.55 [-2.34 to 1.24]

8. Secondary Outcome: The Parkinson's Disease Quality of Life Questionnaire-39 (PDQ-39).
Description: Change from baseline in the Parkinson's Disease Quality of Life Questionnaire-39 (PDQ-39). The PDQ-39 is a self-administered questionnaire of 39 questions relating to 8 key areas of health and daily activities, including both motor and non-motor symptoms. It is scored on a scale of 0 -100 with lower scores indicating better health and high scores indicating more severe symptoms.
Time Frame: Change from Baseline to Week 20
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 40 | 18
score on a scale | -4.88 [-11.46 to 1.69] | -6.29 [-14.81 to 2.23]

9. Secondary Outcome: The Geriatric Depression Scale-15 (GDS-15).
Description: Change from baseline in the Geriatric Depression Scale (GDS-15). The GDS-15 is a 15-item yes/no questionnaire of depression in older adults. Each depressive answer is 1 point. The final score is the tally of the number of depressive answers with the following scores indicating depression: 0-4 No depression; 5-10 Suggestive of a mild depression; 11 + Suggestive of severe depression. The possible scores range from 0 - 15.
Time Frame: Change from Baseline to Week 20
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 41 | 20
score on a scale | 0.30 [-1.30 to 1.89] | 0.27 [-1.74 to 2.27]

10. Secondary Outcome: The Digital Clock Drawing Test (dCDT).
Description: Change from baseline in the digital clock drawing test (dCDT). The pen-like dCDT device will be used to gather the x-y coordinates that describe the movement of the stylus as it changes its position during the assessment. It also assesses when the stylus or writing device is not exerting pressure on the writing surface. The dCDT score is a number from 0 and 100 that represents a person's overall cognitive function as assessed by DCT clock. The total possible score is 100. A negative value of change means a deterioration and a positive value of change means an improvement.
Time Frame: Change from Baseline to Week 20
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 36 | 20
score on a scale | 9.25 [1.69 to 16.80] | 1.58 [-7.61 to 10.77]

11. Secondary Outcome: Power of Attention, Cognitive Reaction Time, and Speed of Memory on the Cognitive Drug Research Computerized Cognition Battery (CDR-CCB) as Assessed by Change From Baseline in CDR-CCB.
Description: The CDR-CCB is an automated cognitive function assessment system. The secondary efficacy outcomes involved the following composite scores:
  * Power of Attention: Min: 350 ms ; Max: 60000 ms
  * Cognitive Reaction Time: Min: - 30000 ms; Max : 30000 ms
  * Speed of Memory: Min 800 ms; Max: 120000 ms
  Higher scores reflect poorer ability, and a positive change from baseline reflects impairment compared to baseline.
Time Frame: Change from Baseline to Week 20
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ms
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 35 | 16
ms
  Power of Attention | 28.14 (90.89) | 133.32 (90.89)
  Cognitive Reaction Time | -49.49 (75.69) | 35.45 (75.69)
  Speed of Memory: number analyzed (Participants) | 33 | 16
  Speed of Memory | 46.97 (331.56) | 232.33 (331.56)

ADVERSE EVENTS:
Time Frame: 24 Months
Arm/Group | GRF6021 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/25
Serious Adverse Events (participants affected / at risk) | 5/51 | 0/25
Other Adverse Events (participants affected / at risk) | 45/51 | 20/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GRF6021 (N=51) | Placebo (N=25)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastritis (General disorders) | 1 (1) | 0 (0)
Mental Changes (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GRF6021 (N=51) | Placebo (N=25)
Headache (Nervous system disorders) | 8 (8) | 2 (2)
Dizziness (Nervous system disorders) | 5 (5) | 1 (1)
Blood pressure diastolic decreased (Investigations) | 2 (2) | 4 (4)
Hypotension (Vascular disorders) | 6 (6) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 7 (7) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement contains language that restricts the PI from discussing or publishing Sponsor confidential and/or proprietary information. The embargo period may be extended by mutual agreement of the Sponsor and PI.

DOCUMENTS (2):
  • Study Protocol (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT03713957/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT03713957/SAP_001.pdf